CLINICAL TRIAL: NCT03867006
Title: Optimization of the Preservation of Muscle Mass and / or Its Recovery by a Protein-energy Chrononutrition Approach Dissociated From Meals
Acronym: CARBOPTIMUS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stop funding by Regional Council of Auvergne-Rhône-Alpes, France
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Bioparhom, France (Unknown); Regional Council of Auvergne-Rhône-Alpes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18CH036; 2018-A00712-53 (Other: ANSM)
Record Dates: First submitted 2018-10-22; First posted 2019-03-07 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Undernutrition
Keywords: Malnutrition; Undernutrition; Elderly; Protein; Carbohydrate
MeSH Terms: conditions — Malnutrition | interventions — Proteins; Carbohydrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (No Intervention): Patients will be randomized in the control group. They will have test MNA (Mini Nutritional Assessment), frailty screening tool (questionnaire FiND), clinical examination, blood sample, blood sample with heparin, white blood cells, urine sample, stool sample, maximal voluntary contraction of quadriceps, walking test, get up-and-go test, Hand Grip test, physical activity questionnaire, bioelectrical impedance analysis and Dual Energy X-ray Absorptiometry (DEXA).
- protein group (Experimental): Patients will be randomized in the protein group. They will have test MNA (Mini Nutritional Assessment), frailty screening tool (questionnaire FiND), clinical examination, blood sample, blood sample with heparin, white blood cells, urine sample, stool sample, maximal voluntary contraction of quadriceps, walking test, get up-and-go test, Hand Grip test, physical activity questionnaire, bioelectrical impedance analysis, Dual Energy X-ray Absorptiometry (DEXA) and protein.
  Interventions: Dietary Supplement: Protein
- protein and carbohydrates group (Experimental): Patients will be randomized in the protein and carbohydrates group. They will have test MNA (Mini Nutritional Assessment), frailty screening tool (questionnaire FiND), clinical examination, blood sample, blood sample with heparin, white blood cells, urine sample, stool sample, maximal voluntary contraction of quadriceps, walking test, get up-and-go test, Hand Grip test, physical activity questionnaire, bioelectrical impedance analysis, Dual Energy X-ray Absorptiometry (DEXA) and protein and carbohydrates.
  Interventions: Dietary Supplement: Protein and Carbohydrate

INTERVENTIONS:
Dietary Supplement: Protein — In addition to their normal meal, patients will eat 30g of whey protein every lunch during 90 days.
  Arms: protein group
Dietary Supplement: Protein and Carbohydrate — In addition to their normal meal, patients will eat 30g of whey protein every lunch during 90 days and eat 60g of carbohydrates 2h after every diner during 90 days.
  Arms: protein and carbohydrates group

SUMMARY:
Muscle wasting has a multifactorial origin, including decreased physical activity, malnutrition, loss of post-incident muscle recovery abilities, and decreased ability to regenerate muscle. Among the strategies tested to improve the production of proteins and thus muscle is the supplementation of whey proteins. However this strategy does not seem sufficient and optimal to avoid muscle wasting and it must be complemented by a complementary action.

Muscle protein degradation also occurs during the nocturnal fasting periods to provide amino acids for energy purposes and to produce glucose, essential for vital organs. The preservation of the benefit of whey intake during meals could therefore be optimized by reducing the use of muscle proteins for energy purposes during the night.

DETAILED DESCRIPTION:
In this study, three arms will be studied for 3 months: 1 control group, 1 group with whey supplementation at lunch, and 1 group with whey supplementation at lunch and an energy bolus before bedtime. Actions include weight and body composition monitoring, nutritional status and muscle function, as well as mechanistic.

ELIGIBILITY:
Inclusion Criteria:

* Resident on the Accommodation Establishments for Dependent Elderly Persons on the Mutuality of Loire, France
* Risk of undernutrition or moderate undernutrition with one of the following criteria :

  * Either 5-10% of weight loss in 1 month or 10-15% in 6 months.
  * Or Body Mass Index (BMI) between 16 and 21
  * Or Albumin levels between 30 and 35 g/L
  * Or global Mini Nutritional Assessment (MNA) test between 17 and 23.5
  * Or Short Emergency Geriatric Assessment (SEGA) Score >8

Exclusion Criteria:

* Sub-acute pathology (flu, gastroenteritis, bacterial infections ...) or trauma (fracture, surgery ...) in the 30 days prior to inclusion.
* Hepatocellular insufficiency
* Heart failure with decompensation
* Severe dementia,
* Insulin-treated diabetes
* Renal insufficiency (clearance <30 ml / min)
* Long-term cortico-therapy
* Cancer undergoing chemotherapy treatment or/and radiotherapy
* Gastrointestinal pathology,
* Diet incompatible with the nutritional protocol (intolerance to milk or lactose, vegetarians, vegans, ...)
* Motor disability leading to the impossibility of doing muscle function tests.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Appendicular lean body mass (gramme) | Days 0 and 90
  Comparison appendicular lean body mass between the day of inclusion and 90 days after. It is measuring by Dual Energy X-ray Absorptiometry (DEXA).

SECONDARY OUTCOMES:
total body composition | Days 0, 45 and 90
  Correlation between Dual Energy X-ray Absorptiometry (DEXA) results and bioelectrical impedance analysis results to determine total body composition.
Plasma albumin level (g/l) | Days 0, 45 and 90
  blood sample.
Frailty screening tool | Days 0 and 90
  Determination of fragility status. 3 status : Dependent, Fragile, Robust
Mini Nutritional Assessment score | Days 0 and 90
  Determine nutritional status. Score : 0-30
Inflammatory status | Days 0, 45 and 90
  Analysis of inflammatory status by blood sample results. C-reactive protein (CRP), Interleukin 6 (IL-6), Tumor necrosis factor (TNFα), monocyte chemoattractant protein 1 (MCP1)
Hand Grip test (N) | Days 0 and 90
  Analysis of muscle function tests.
6 minutes walk test (m) | Days 0 and 90
  Analysis of muscle function tests.
Maximal voluntary contraction of quadriceps (N) | Days 0 and 90
  Analysis of muscle function tests.
Get up-and-go test (s) | Days 0 and 90
  Analysis of muscle function tests.
Profiles of the differential expression of potentials biomarkers | Days 0, 45 and 90
  Analysis of profiles of the differential expression of potentials biomarkers by results of blood sample with heparin, urine sample and white blood cells.
microbiota | Days 0 and 90
  Analysis of microbiota by stool sample results.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio POLAKOF, PhD, Study Director — UMR 1019, INRA, France
Locations (3):
- France (3):
  - EHPAD Cité des Aînés, Saint-Etienne
  - EHPAD La Cerisaie, Saint-Etienne
  - EHPAD Le Soleil, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No